CLINICAL TRIAL: NCT03157778
Title: Relation Between Pregnenolone Endocannabinoids in Normal-weight and Obese Men
Acronym: CannaPREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/33
Record Dates: First submitted 2017-05-05; First posted 2017-05-17 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: pregnenolone; endocannabinoid; food intake; type-1 cannabinoid receptor
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Obese men versus normal-weight men
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese men (Experimental): Measured plasmatic concentration of pregnenolone and endocannabinoid in fasting conditions and over a meal in obese men.
  Interventions: Other: Obese men
- Normal-weight men (Active Comparator): Measured plasmatic concentration of pregnenolone and endocannabinoid in fasting conditions and over a meal in normal-weight men.
  Interventions: Other: Normal-weight men

INTERVENTIONS:
Other: Obese men — Biological measures before, just before, and after lunch, in obese men
  Arms: Obese men
Other: Normal-weight men — Biological measures before, just before, and after lunch, in normal-weight men.
  Arms: Normal-weight men

SUMMARY:
Measured plasmatic concentration of pregnenolone and endocannabinoid in fasting conditions and over a meal in obese and normal-weight men subjects, to research a dysfunction in the negative feed-back between pregnenolone and CB1 ligand in obese subjects. This dysfunction could participate to the hyperactivity of endocannabinoid system saw in obesity.

DETAILED DESCRIPTION:
Endocannabinoid system is an orexigenic key system, controlling the energy balance. It is composed of receptors (ex: CB1), of endogenous ligands, the endocannabinoids (ex: anandamide and 2- arachidonoylglycerol) and of enzymes implied in the synthesis and the degradation of the endocannabinoids. Researches resulting from our group highlighted anomalies of the plasmatic concentrations of endocannabinoid, in obese subject compared to normal-weight subject. Those being higher in obese subject with a flatness of post prandial reduction of AEA, so maintenance of elevated levels which can facilitate the food catch and create a metabolic vicious circle. In addition, prestigious research resulting from our collaborators highlighted in the animal that exposure to tetrahydrocannabinol (THC, ligand exogenic of CB1) induced the synthesis of pregnenolone (neurosteroid) which, by an autocrine effect on the CB1, inhibited the effects of the THC. In particular one of the principal behavioural effects: the food intake.

We want to measure pregnenolone and endocannabinoid concentrations in men blood samples, to observe if this association exists in fasting conditions and over a meal in normal-weight and obese subjects. Obese subjects will be recruited during an hospitalization, while normal subject will be recruited by a poster at Bordeaux university and Haut-Leveque hospital. They will be included at Haut-Leveque hospital during morning at hospital.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects:

  * men,
  * aged between 18 and 65 years,
  * BMI>30kg/m2.
* Normal-weight subjects:

  * men,
  * aged between 18 and 65 years,
  * BMI<25kg/m2.

Exclusion Criteria:

* For all subjects:

  * cannabis detected by urinary tetrahydrocannabinol presence,
  * treatment which can interfere with endocannabinoid system (antidepressant, antipsychotics, anxiolytics).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Comparison of pregnenolon plasmatic concentration in both groups. | Change from 1 hour before lunch to 1 hour after lunch at inclusion day
  Pregnenolon plasmatic concentration will be measured at several points.

SECONDARY OUTCOMES:
Comparison of neurosteroid plasma concentrations and endocannabinoid plasma concentrations | Change from 1 hour before lunch to 1 hour after lunch at inclusion day
  Neurosteroid and endocannabinoid plasma concentrations will be measured at several points.
Comparison of endocannabinoid plasma concentration and pregnenolone plasma concentration | Change from 1 hour before lunch to 1 hour after lunch at inclusion day
  Endocannabinoid and pregnenolone concentrations will be measured at several points.

CONTACTS AND LOCATIONS:
Overall Officials: Lhomme Edouard, Dr, Study Chair — USMR
Locations (1):
- Hôpital Haut-Lévêque, Pessac, France

IPD SHARING:
Plan to Share IPD: No